CLINICAL TRIAL: NCT01391221
Title: Inflammatory Markers and Cognitive Function in Major Depression:a Pilot Study
Brief Title: Inflammatory Markers and Cognitive Function in Major Depression
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre de Recherche de l'Institut Universitaire en santé Mentale de Montréal (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Smadar Valerie Tourjman, MDCM, FRCPc, MSc, Centre de Recherche de l'Institut Universitaire en santé Mentale de Montréal
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2011005
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2011-07

CONDITIONS: Major Depression
Keywords: Depression; Inflammation; Cognition; Pain; Allostatic load
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Inflammation; Pain | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Duloxetine treatment (Experimental): Subjects with major depression will be entered into the trial and treated with open label duloxetine
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — Subjects with major depression will be entered into the trial and treated with duloxetine 30 mg for one week, followed by 60 mg for 8 weeks. The option of increasing the dose as clinically indicated to 120mg is possible for the last 4 weeks of the study intervention
  Other Names: Cymbalta

SUMMARY:
Major depression is accompanied by cognitive changes as well as alterations in multiple physical functions. The inflammatory system is altered generally toward a pro-inflammatory state. Antidepressants are associated with a decrease in this proinflammatory state. This study aims to generate pilot data concerning a possible link between cognition, inflammation and response to treatment. The cognitive function of subjects with major depression will be tested before and after treatment with duloxetine. Inflammatory markers will be measured at both time points.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-50 Primary diagnosis of major depression Ability to give informed consent

Exclusion Criteria:

* Neurologic disorders affecting cognition
* Unstable or untreated medical disorders
* Medical disorders associated with pain
* Recent pregnancy or delivery
* Psychiatric disorders other than MD which are the primary focus of treatment
* Treatment with antidepressants in the past 4 weeks

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Cognitive function measured by CANTAB | 12 weeks
  Correlation between cytokines and cognitive function

SECONDARY OUTCOMES:
pain inhibition | 12 weeks
  Correlation between depression, antidepressant treatment status, inflammation and inhibition of perception of pain stimulus
Allostatic load | 12 weeks
  Correlation between depressive symptoms, antidepressant treatment status and allostatic load

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Centre de Recherche Fernand Seguin, Montreal, Quebec
  - Hôpital Maisonneuve Rosemont, Montreal, Quebec